CLINICAL TRIAL: NCT02044848
Title: A Randomized, Double-blind, Multiple Dose, Placebo-controlled Study to Evaluate the Safety, Tolerability, Immunogenicity, Pharmacokinetics, and Efficacy of Secukinumab in Adult and Pediatric Patients With New-onset Type 1 Diabetes Mellitus(T1D)
Brief Title: Study of Secukinumab in Patients With Newly-diagnosed Type 1 Diabetes Mellitus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated prematurely by the Sponsor for business reasons only.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAIN457A2227
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Results first posted 2015-10-09 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-01

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: type 1 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Secukinumab (Experimental): Secukinumab will be delivered as part of an induction regimen followed by a maintenance regimen for up to 1 year
  Interventions: Drug: Secukinumab
- Placebo (Placebo Comparator): Placebo will be delivered as part of an induction regimen followed by a maintenance regimen for up to 1 year
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Secukinumab
  Arms: Secukinumab
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study will assess the safety and efficacy of secukinumab on the preservation of pancreatic beta cells in patients with newly-diagnosed type 1 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

Males and females aged 18-35 years initially (subjects aged 8-17 may be included at a later stage, starting with age 12-17 years, followed by age 8-11 years).

Body weight between 40-120 kg initially (subjects weighing 21-39 kg may be included at a later stage).

Recent onset type 1 diabetes mellitus, diagnosed with 100 days of first dose. Peak stimulated C-peptide levels >/= 0.2 pmol/L following mixed meal tolerance test

Exclusion Criteria:

Any form of diabetes other than auto-immune type 1 (eg, type 2 diabetes, maturity onset diabetes of the young, latent autoimmune diabetes of the adult).

Diabetic ketoacidosis within 2 weeks of screening. Pregnancy or lactation. Recent (within 2 weeks of screening), ongoing, chronic or recurrent infectious disease.

Active infection with hepatitis B or C, Epstein-Barr virus, cytomegalovirus, or HIV.

Tuberculosis infection. Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2014-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- United States (2):
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only adult patients were enrolled (no pediatrics as planned) and no one completed the planned treatment period.
Period: Overall Study
Arm/Group | Secukinumab | Placebo
Started | 2 | 3
Completed | 0 | 0
Not Completed | 2 | 3
Not completed — Administrative Problems | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab | Placebo | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 24 (4.24) | 24 (1.73) | 24 (2.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Stimulated C-peptide in Response to a Standard Mixed Meal Tolerance Test
Description: Study was terminated and no data were collected for the Outcome Measure.
Time Frame: Week 52
Population: Study was terminated and no data were collected for the Outcome Measure
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Secukinumab | Placebo
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 2/2 | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab (N=2) | Placebo (N=3)
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Blood ketone body (Investigations) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.